CLINICAL TRIAL: NCT03023891
Title: Pharmacogenomics of the Variability in the In Vivo Response to Glucocorticoids
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Vivian Kawai, Research Assistant Professor, Vanderbilt University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 161942; 5K23GM117395-03 (NIH)
Record Dates: First submitted 2017-01-12; First posted 2017-01-18 (Estimated); Results first posted 2020-01-06 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-05

CONDITIONS: Glucocorticoids Toxicity; Glucose Intolerance
Keywords: glucocorticoids; efficacy; metabolic toxicity
MeSH Terms: conditions — Glucose Intolerance | interventions — Prednisone; Drugs, Generic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Prednisone (Experimental): Each participant will received a single dose of oral 60 mg of prednisone
  Visit 1: Baseline Oral Glucose Tolerance Test (OGTT) and White Blood Count (WBC) count Visit 2: Prednisone 60mg oral at 7am, OGGT and WBC count at 4 to 8 hours post drug
  Interventions: Drug: Prednisone

INTERVENTIONS:
Drug: Prednisone — Prednisone 60 mg tablet once
  Other Names: generic, not applicable

SUMMARY:
This study evaluates the effect of acute administration of oral prednisone in white blood cells counts and glucose tolerance and the relationship of these measures with changes in gene expression in healthy volunteers. White blood cells counts, glucose tolerance and gene expression will be study before and after prednisone administration.

DETAILED DESCRIPTION:
Prednisone is a potent anti-inflammatory drug that has large variability in its response. The large inter individual variability in the response to prednisone has a genetic component, but the genetic determinants of this variability remain unknown. We propose to use two relevant phenotypes, changes in white blood cell counts and changes in glucose tolerance induced by in vivo administration of prednisone, to characterize gene expression patterns and identify variants that are involved in the in vivo response to prednisone.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 45 years old (to exclude the effect of age on glucose tolerance);
* BMI between 20 and 25 kg/m2 (to exclude individuals that are likely to have impaired insulin response);
* Normal fasting glucose;
* Stable weight for three months before participation

Exclusion Criteria:

* BMI >25kg/m2;
* Fasting glucose ≥126 mg/dl
* Shift work or disordered sleep (to exclude individuals with alterations in the hypothalamus-adrenergic axis);
* Any diseases;
* Use of any medication regularly (including over-the-counter);
* Previous exposure to glucocorticoids (within the last year);
* Pregnancy

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2017-02-15 (Actual); Primary Completion 2019-01-10 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vivian K Kawai, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center -CRC, Nashville, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 25 participants signed consent, 5 did not show up for screening and 2 failed screening. 18 participants started the study.
Groups:
- Prednisone: Each participant will received a single dose of oral 60 mg of prednisone
  Prednisone: Prednisone 60 mg tablet once
Period: Overall Study
Arm/Group | Prednisone
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Prednisone
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 14
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: White Blood Cell Counts
Description: White Blood Count at baseline (Visit 1) and within 4 to 8 hours after drug administration (Visit 2)
Time Frame: baseline and within 4 and 8 hours after drug administration
Measure: Mean (Standard Deviation); unit: x10^3 cells/mL
Arm/Group | Prednisone
Number analyzed (Participants) | 18
x10^3 cells/mL
  Visit 1: baseline | 5.26 (0.92)
  Visit 2: 4 to 8 hours post prednisone | 6.99 (1.39)

2. Primary Outcome: Glucose Tolerance Test: Area Under the Curve (AUC) for Plasma Glucose
Description: AUC for plasma glucose during glucose tolerance test at baseline and 4-8 hours after drug administration.
  Plasma glucose levels were measured at 0, 10, 20, 30, 60, 90 and 120 minutes during glucose tolerance test at baseline (Visit 1) and after drug administration (Visit 2)
Time Frame: baseline and 4-8 hours after drug administration
Measure: Mean (Standard Deviation); unit: mg*min/dL
Arm/Group | Prednisone
Number analyzed (Participants) | 18
mg*min/dL
  Visit 1: baseline | 13530.56 (2002.23)
  Visit 2: 4-8 hours post prednisone | 20273.75 (3973.26)

3. Primary Outcome: Glucose Tolerance Test: Area Under the Curve (AUC) for Insulin Levels
Description: AUC for insulin levels during glucose tolerance test at baseline and 4-8 hours after prednisone.
  Insulin levels were measured at 0, 10, 20, 30, 60, 90 and 120 minutes during glucose tolerance test at baseline (Visit 1) and after drug administration administration (Visit 2).
Time Frame: baseline and 4-8 hours after drug administration
Measure: Mean (Standard Deviation); unit: μU*min/mL
Arm/Group | Prednisone
Number analyzed (Participants) | 18
μU*min/mL
  Visit 1: baseline | 5415.87 (2344.63)
  Visit 2: 4-8 hours post prednisone | 5466.55 (2382.49)

4. Primary Outcome: Glucose Tolerance Test: Area Under the Curve (AUC) for C-peptide Levels
Description: AUC for C-peptide during glucose tolerance test at baseline and 4-8 hours after prednisone.
  C-peptide levels were measured at 0, 10, 20, 30, 60, 90, and 120 minutes during glucose tolerance test at baseline (Visit 1) and after drug administration (Visit 2)
Time Frame: baseline and 4-8 hours after drug administration
Measure: Mean (Standard Deviation); unit: ng*min/mL
Arm/Group | Prednisone
Number analyzed (Participants) | 18
ng*min/mL
  Visit 1: baseline | 493.89 (135.77)
  Visit 2: 4-8 hours post prednisone | 449.41 (101.27)

ADVERSE EVENTS:
Time Frame: 2 days
Groups:
- Prednisone: Each participant will received a single dose of oral 60 mg of prednisone
  Visit 1: Baseline Oral Glucose Tolerance Test (OGTT) and White Blood Count (WBC) count Visit 2: Prednisone 60 mg oral at 7am, OGGT and WBC count at 4 to 8 hours post drug
  Prednisone: Prednisone 60 mg tablet once
Arm/Group | Prednisone
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 4/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prednisone (N=18)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Mild Dizziness (General disorders) | 1 (1)
Mild anxiety and hyperactivity (General disorders) | 1 (1)
Tiredness, Fatigue (General disorders) | 1 (1)
Dehydration (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2018-10-31): https://cdn.clinicaltrials.gov/large-docs/91/NCT03023891/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2017-10-23): https://cdn.clinicaltrials.gov/large-docs/91/NCT03023891/Prot_SAP_001.pdf